CLINICAL TRIAL: NCT05167149
Title: A Randomized Controlled Comparison Study of Carbon Nanoparticles and Indocyanine Green for Sentinel Lymph Node Biopsy in Early Stage Cervical Cancer
Brief Title: Carbon Nanoparticles and Indocyanine Green for Sentinel Lymph Node Biopsy in Early Stage Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CFH2020-2-4024
Record Dates: First submitted 2021-01-15; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-01

CONDITIONS: Cervical Cancer Stage IB1
Keywords: Early Stage Cervical Cancer; Sentinel Lymph Node Biopsy; Carbon Nanoparticle; Indocyanine Green; Ultrastaging
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon nanoparticles group (Experimental)
  Interventions: Procedure: Carbon nanoparticles
- Indocyanine green group (Active Comparator)
  Interventions: Procedure: Indocyanine green

INTERVENTIONS:
Procedure: Carbon nanoparticles — After pneumoperitoneum is established and laparoscopic instruments are prepared, according to National Comprehensive Cancer Network (NCCN) guidelines, 1ml diluted ICG solution (25 mg /10 ml) is injected into the submucosa around tumor at 3 and 9 o'clock of the cervix (2ml totally) with 1ml syringe. ICG should be slowly injected to avoid drug leakage. Intratumoral and deep cervical stroma injection should be avoided. The retroperitoneum is dissected immediately after injection under the multimodel observation of fluorescence laparoscopy. Search the fluorescent labeled lymphatics from bilateral parametrium to iliac vessels. The diffusion of ICG is rapid , and it is easy to spread to the next stations lymph nodes. The first fluorescent labeled lymph nodes on each lymphatic drainage pathway are identified as SLNs, other than all fluorescent lymph nodes. All detectable SLNs and enlarged or suspicious nodes regardless of mapping are resected for pathological examination alone.
  Arms: Carbon nanoparticles group
Procedure: Indocyanine green — After pneumoperitoneum is established and laparoscopic instruments are prepared, according to NCCN guidelines, 0.5ml(25mg) carbon nanoparticle solution (the dose was from our retrospective study) is injected into the submucosa around tumor at 3 and 9 o'clock of the cervix (1ml totally) with 1ml syringe. Carbon nanoparticle should be slowly injected to avoid drug leakage. Intratumoral and deep cervical stroma injection should be avoided. The retroperitoneum is dissected immediately after injection. Search the black lymphatics from bilateral parametrium to iliac vessels. Because there is no fluorescence penetration as ICG, the black lymphatic vessels should be dissected carefully.The first black lymph nodes on each lymphatic drainage pathway are identified as SLNs, other than all black lymph nodes. All detectable SLNs and enlarged or suspicious nodes regardless of mapping are resected for pathological examination alone.
  Arms: Indocyanine green group

SUMMARY:
The metastasis rate of pelvic lymph node in early cervical cancer is low. Systemic lymph node resection is traumatic and has many complications. Sentinel lymph node (SLN) biopsy can effectively avoid unnecessary lymph node dissection, which has been recommended in clinical guidelines. Indocyanine green(ICG) fluorescence imaging as the method of SLN mapping is recommended in international guidelines. However, the imaging equipment is very expensive which limits the popularization of ICG in different medical centers of various surgical volumes. Carbon nanoparticle is an innovative tracer without any special imaging equipment for SLN mapping in China. Some retrospective researches have proved that carbon nanoparticle is effective, simple, economic and suitable for popularization in different medical centers. In this study, a prospective randomized controlled trial will be conducted to analyze the non-inferiority of carbon nanoparticles compared to ICG, and to verify the application value of carbon nanoparticles. 144 cervical cancer patients with stage IB1 (FIGO2018) will be prospectively enrolled and randomly divided into two groups (R = 1:1). 72 patients will undergo SLN biopsy with carbon nanoparticles and 72 patients will be mapped by ICG. The primary endpoint is overall SLN detection rate. The secondary endpoints include bilateral SLN detection rate, the number of SLN detected, sensitivity, false negative rate and negative predictive value of SLN biopsy. Diagnostic accuracy will be evaluated at both pelvis and patient levels. What's more, SLN pathological ultrastaging will be conducted to increase the diagnostic accuracy. The hypothesis of this study is that the overall SLN detection rate by carbon nanoparticles is not inferior to that using ICG. And the differences of bilateral SLN detection rate, sensitivity, false negative rate and negative predictive value between two groups are not significant.

DETAILED DESCRIPTION:
This is a prospective randomized controlled non-inferiority trial. Patients with early stage cervical cancer who met the inclusion criteria are divided into carbon nanoparticle group and ICG group by block random method. It is assumed that the overall SLN detection rate was PT (90%) in experimental group(carbon nanoparticle) and was PC (85%) in control group (ICG). The non-inferiority threshold Δ is -10%. The type I error and type II error of the hypothesis test are set as 0.05 and 0.2 respectively. The sample size is 60 cases in each group calculated by"Non inferiority tests for two proportions"method of Power Analysis and Sample Size (PASS) Software 11.0. After calculation, considering the 20% shedding rate, the sample size is 144 totally. There are 72 cases in experimental group and 72 cases in control group. Radical hysterectomy and systemic pelvic lymph node dissection are conducted after SLN resection, and paraaortic lymph node biopsy is conducted when necessary. Sentinel lymph nodes will be cut at 2-mm intervals perpendicular to the long axis in a bread-loaf fashion. Sentinel lymph nodes are then fixed in formalin and embedded in paraffin. Routine hemotoxin & eosin(H&E) staining is used for each SLN. Subsequent ultrastaging is performed if the initial H&E assessment is negative. SLN ultrastaging is performed by cutting three 5-μm sections at two levels, 50-μm apart, from each paraffin block of negative SLN. At the first level, two adjacent 5-μm sections are stained with H&E and immuno-histochemistry using the anti-cytokeratin AE1:AE3, respectively. At the second level, one 5-μm section is evaluated by H&E staining. Nonsentinel lymph nodes are bisected parallel to the long axis and stained with H&E staining.Nodal metastases are classified as (1) isolated tumor cells (ITCs) (single cells or clusters ≤ 0.2mm in largest dimension),(2) micrometastases (tumor deposits 0.2mm-2 mm), or (3) macrometastases (tumor deposits > 2mm). All pathological reviews will be finished by two independent gynecologic pathologists in the Department of Pathology of Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College. A third senior pathologist is invited to decide the diagnosis when discordance occurs.

ELIGIBILITY:
Inclusion Criteria:

* Cervical squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma diagnosed by pathological biopsy;
* Tumor stage is IB1 (FIGO 2018);
* No distant metastasis (chest, abdominal and pelvic enhanced CT or positron emission tomography (PET) -CT);
* 18-70 years old;
* Eastern Cooperative Oncology Group (ECOG) score ≤ 2 and tolerable for radical hysterectomy and systemic lymph node resection;
* No obvious dysfunction or chronic disease of heart, liver and kidney, and no history of other malignant tumors;
* Volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Residual cervical cancer;
* Small cell carcinoma, neuroendocrine carcinoma and other special histological types;
* Patients who have received radiotherapy or chemotherapy before enrollment;
* Allergic constitution, allergic to iodine;
* ICG skin test is positive;
* Patients considered unsuitable for inclusion by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Overall SLN detection rate | From date of operation to the date of completion of routine pathological examination, usually 2 weeks after operation.
  The percentage of patients with successfully detected SLNs in all eligible patients.

SECONDARY OUTCOMES:
Bilateral SLN detection rate | From date of operation to the date of completion of routine pathological examination, usually 2 weeks after operation.
  The percentage of patients with successfully detected SLNs in both sides of the pelvis in all eligible patients
The number of detected SLNs | From date of operation to the date of completion of routine pathological examination, usually 2 weeks after operation.
  The numbers of detected SLNs are calculated by the pathologist.
Location of SLNs | From date of operation to the date of completion of routine pathological examination, usually 2 weeks after operation.
  Distribution of SLNs in pelvic and abdominal cavity, including external iliac, obturator fossa, internal ilia, deep inguinal, common iliac, presacral, inferior vena cava, para-aortic, and parametrial regions.
Sensitivity of SLN biopsy | From date of operation to the date of completion of SLNs pathological ultrastaging. 3 years.
  The percentage of patients or pelvises with positive SLNs in pathological examination among those with positive pelvic lymph nodes.
False negative rate | From date of operation to the date of completion of SLNs pathological ultrastaging. 3 years.
  The percentage of patients or pelvises with negative SLNs in pathological examination among those with positive pelvic lymph nodes.
Negative predictive value | From date of operation to the date of completion of SLNs pathological ultrastaging. 3 years.
  The percentage of patients or pelvises with negative pelvic lymph nodes among those whose SLNs were negative in pathological examination.

OTHER OUTCOMES:
Duration of operation | One month.
  The time from the beginning of the operation to the end of the operation.
Intraoperative bleeding volume | One month.
  The amount of bleeding during the operation.
Adverse events caused by injection of tracers. | From the time of tracer injection to the date of leaving hospital.
  Adverse events, such as allergy, are caused by injection of tracers and defined according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Operative complications | From the beginning of operation to 6 months after operation.
  In this study, operative complications are defined according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, M.D., Study Chair — Department of Gynecological Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Gynecological Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Cibula D, Dusek J, Jarkovsky J, Dundr P, Querleu D, van der Zee A, Kucukmetin A, Kocian R. A prospective multicenter trial on sentinel lymph node biopsy in patients with early-stage cervical cancer (SENTIX). Int J Gynecol Cancer. 2019 Jan;29(1):212-215. doi: 10.1136/ijgc-2018-000010. PMID 30640706
- [Background] Cibula D, McCluggage WG. Sentinel lymph node (SLN) concept in cervical cancer: Current limitations and unanswered questions. Gynecol Oncol. 2019 Jan;152(1):202-207. doi: 10.1016/j.ygyno.2018.10.007. Epub 2018 Oct 11. PMID 30318103
- [Background] Frumovitz M, Plante M, Lee PS, Sandadi S, Lilja JF, Escobar PF, Gien LT, Urbauer DL, Abu-Rustum NR. Near-infrared fluorescence for detection of sentinel lymph nodes in women with cervical and uterine cancers (FILM): a randomised, phase 3, multicentre, non-inferiority trial. Lancet Oncol. 2018 Oct;19(10):1394-1403. doi: 10.1016/S1470-2045(18)30448-0. Epub 2018 Aug 22. PMID 30143441
- [Background] Salvo G, Ramirez PT, Levenback CF, Munsell MF, Euscher ED, Soliman PT, Frumovitz M. Sensitivity and negative predictive value for sentinel lymph node biopsy in women with early-stage cervical cancer. Gynecol Oncol. 2017 Apr;145(1):96-101. doi: 10.1016/j.ygyno.2017.02.005. Epub 2017 Feb 8. PMID 28188015
- [Background] Buda A, Crivellaro C, Elisei F, Di Martino G, Guerra L, De Ponti E, Cuzzocrea M, Giuliani D, Sina F, Magni S, Landoni C, Milani R. Impact of Indocyanine Green for Sentinel Lymph Node Mapping in Early Stage Endometrial and Cervical Cancer: Comparison with Conventional Radiotracer (99m)Tc and/or Blue Dye. Ann Surg Oncol. 2016 Jul;23(7):2183-91. doi: 10.1245/s10434-015-5022-1. Epub 2015 Dec 29. PMID 26714944
- [Background] Bats AS, Frati A, Mathevet P, Orliaguet I, Querleu D, Zerdoud S, Leblanc E, Gauthier H, Uzan C, Deandreis D, Darai E, Kerrou K, Marret H, Lenain E, Froissart M, Lecuru F. Contribution of lymphoscintigraphy to intraoperative sentinel lymph node detection in early cervical cancer: Analysis of the prospective multicenter SENTICOL cohort. Gynecol Oncol. 2015 May;137(2):264-9. doi: 10.1016/j.ygyno.2015.02.018. Epub 2015 Feb 26. PMID 25727652
- [Background] Imboden S, Papadia A, Nauwerk M, McKinnon B, Kollmann Z, Mohr S, Lanz S, Mueller MD. A Comparison of Radiocolloid and Indocyanine Green Fluorescence Imaging, Sentinel Lymph Node Mapping in Patients with Cervical Cancer Undergoing Laparoscopic Surgery. Ann Surg Oncol. 2015 Dec;22(13):4198-203. doi: 10.1245/s10434-015-4701-2. Epub 2015 Jun 30. PMID 26122376
- [Background] Zuo J, Wu LY, Cheng M, Bai P, Lei CZ, Li N, Zhang GY, Zhao D, Li B. Comparison Study of Laparoscopic Sentinel Lymph Node Mapping in Endometrial Carcinoma Using Carbon Nanoparticles and Lymphatic Pathway Verification. J Minim Invasive Gynecol. 2019 Sep-Oct;26(6):1125-1132. doi: 10.1016/j.jmig.2018.11.002. Epub 2018 Nov 14. PMID 30445188
- [Background] Kim CH, Soslow RA, Park KJ, Barber EL, Khoury-Collado F, Barlin JN, Sonoda Y, Hensley ML, Barakat RR, Abu-Rustum NR. Pathologic ultrastaging improves micrometastasis detection in sentinel lymph nodes during endometrial cancer staging. Int J Gynecol Cancer. 2013 Jun;23(5):964-70. doi: 10.1097/IGC.0b013e3182954da8. PMID 23694985
- [Background] Cusimano MC, Vicus D, Pulman K, Maganti M, Bernardini MQ, Bouchard-Fortier G, Laframboise S, May T, Hogen LF, Covens AL, Gien LT, Kupets R, Rouzbahman M, Clarke BA, Mirkovic J, Cesari M, Turashvili G, Zia A, Ene GEV, Ferguson SE. Assessment of Sentinel Lymph Node Biopsy vs Lymphadenectomy for Intermediate- and High-Grade Endometrial Cancer Staging. JAMA Surg. 2021 Feb 1;156(2):157-164. doi: 10.1001/jamasurg.2020.5060. PMID 33175109
- See also: Clinical analysis of 76 cases of sentinel lymph node detection in cervical cancer and endometrial cancer — http://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDZHYX&filename=ZHFC201709010&v=gM0%25mmd2F6%25mmd2FM3JtuIfoz3mZtUhUsBF9Gwt868LTu7I5drBVtlqV7U3suzOW%25mmd2Fw6PsbLgPc